CLINICAL TRIAL: NCT03511586
Title: Total Shoulder Arthroplasty Multi-Center Registry
Status: Recruiting | Type: Observational
Sponsor: Arthrex, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 608
Record Dates: First submitted 2018-04-12; First posted 2018-04-30 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-06

CONDITIONS: Shoulder Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

SUMMARY:
The objective of the study is a multi-center prospective registry to collect clinical outcomes of anatomic and reverse total shoulder arthroplasty.

DETAILED DESCRIPTION:
The study is a non-randomized multi-center prospective registry and subjects will be treated according to standard of care at each center. Subjects will be approached for participation in this study after they have made the decision to undergo a primary or revision shoulder arthroplasty procedure. The treating surgeon will obtain verbal consent from the patient for a research coordinator to screen for eligibility. Patients who meet all criteria will be offered enrollment into the study. The total enrollment goal is a minimum of 500 anatomic shoulder arthroplasty and 500 reverse shoulder arthroplasty subjects enrolled in the multi-center registry.

ELIGIBILITY:
Inclusion Criteria:

1. Patient voluntarily consents to participate in the study and has the mental and physical ability to participate in the study, fill out subjective questionnaires, return for follow-up visits, and comply with prescribed post-operative physical therapy.
2. Patient is between the ages of 18 and 100 years.
3. The patient has a planned primary or revision implantation of an anatomic (hemi-arthroplasty or total arthroplasty) or a reverse shoulder prosthesis system manufactured by Arthrex.
4. Patient has a standard of care preoperative CT taken within 6 months that has been submitted for Arthrex VIP (Virtual Implant Positioning) planning.

Exclusion Criteria

1. Patient has known intentions, obligations, or co-morbidity that would inhibit them from participating in the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients who are seeking treatment or are undergoing a shoulder replacement procedure utilizing an Arthrex shoulder arthroplasty prostheses are being invited to participate in this research registry.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2015-07-28 (Actual); Primary Completion 2035-07 (Estimated); Study Completion 2035-11 (Estimated)

PRIMARY OUTCOMES:
Change in Pain | 10 years
  Measure of pain intensity. This is done with the Visual Analog Scare. (VAS)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (22):
  - University of Arizona/Banner Health, Phoenix, Arizona
  - Banner Medical Group, Phoenix, Arizona
  - Scottsdale, Arizona
  - Denver, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - Andrews Research & Education Foundation, Gulf Breeze, Florida
  - Advent Health Orlando, Orlando, Florida
  - NorthShore University Health System, Evanston, Illinois
  - The Trustees of Indiana University, Indianapolis, Indiana
  - The University of Michigan, Ann Arbor, Michigan
  - Grand Rapids, Michigan
  - Columbia, Missouri
  - The Rothman Institute, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Cleveland Shoulder Institute, Beachwood, Ohio
  - Medford, Oregon
  - Rothman Orthopaedic Institute, Philadelphia, Pennsylvania
  - The Hawkins Foundation, Greenville, South Carolina
  - Germantown, Tennessee
  - University of Virginia, Charlottesville, Virginia
  - Virginia Beach, Virginia
- Orthopädische Chirurgie München (OCM), München, Germany
- Schulthess Klinik, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No